CLINICAL TRIAL: NCT06739512
Title: Efficacy and Safety of Pulsed Field Ablation in Three Different Substrate Ablation Strategies for Persistent Atrial Fibrillation: a Multicenter Randomized Controlled Trial
Brief Title: Pulsed Field Ablation in Three Different Substrate Ablation Strategies for Persistent Atrial Fibrillation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Albert Einstein College of Medicine and Montefiore Medical Center (Unknown); Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine (Unknown); Shandong University of Traditional Chinese Medicine (Other); Yuhuan Second People's Hospital (Unknown); Changshu Hospital of Traditional Chinese Medicine (Other); Jinan People's Hospital (Unknown); Xuzhou Central Hospital (Other); The PLA Navy Anqing Hospital (Unknown)
Responsible Party: Principal Investigator, Xu Liu, MD, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXT-II
Record Dates: First submitted 2024-11-24; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation (AF)
Keywords: ablation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anatomical Guided Ablation Group (Placebo Comparator): This group will undergo pulmonary vein isolation (PVI) combined with anatomical linear ablation based on predefined anatomical landmarks (a complete posterior wall box isolation to ensure comprehensive atrial substrate modification), including lines such as the mitral isthmus and roofline. The ablation will aim to create bidirectional block without relying on electrogram-based mapping.
  Interventions: Procedure: Anatomical Guided Ablation
- Electrogram Guided Ablation Group (Active Comparator): This group will undergo PVI and targeted ablation of atrial fibrillation "drivers" identified through electrogram-guided mapping. The mapping will focus on electrograms with characteristics such as spatial-temporal dispersion, high-frequency potentials, and short local cycle lengths.
  Interventions: Procedure: Electrogram Guided Ablation
- Extensive Electro-Anatomical Guided Ablation Group (Experimental): This group will receive PVI and a combination of anatomical linear ablation (a complete posterior wall box isolation to ensure comprehensive atrial substrate modification) and electrogram-guided ablation. It represents an extensive strategy that integrates both anatomical and potential-based mapping for optimized ablation targeting.
  Interventions: Procedure: Extensive Electro-Anatomical Guided Ablation

INTERVENTIONS:
Procedure: Extensive Electro-Anatomical Guided Ablation — Ablation using PFA. Combination of anatomical and electrogram-guided ablation techniques.
  Arms: Extensive Electro-Anatomical Guided Ablation Group
Procedure: Anatomical Guided Ablation — Ablation using PFA. Guided by anatomical landmarks without potential mapping
  Arms: Anatomical Guided Ablation Group
Procedure: Electrogram Guided Ablation — Ablation using PFA. Guided by real-time electrogram characteristics from a multi-electrode catheter.
  Arms: Electrogram Guided Ablation Group

SUMMARY:
This multicenter, randomized, controlled trial aims to evaluate the efficacy and safety of pulsed field ablation (PFA) in patients with persistent atrial fibrillation (PeAF). We will compare three distinct substrate ablation strategies: anatomical guided ablation (ANAT group), electrogram guided ablation (EGM group), and extensive electro-anatomical guided ablation (EXT group). The study seeks to identify which ablation strategy yields the highest efficacy and safety profiles to potentially guide future clinical practice in the management of PeAF.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-80 years diagnosed with persistent atrial fibrillation.
2. Ineffectiveness or intolerance to at least one Class I or III anti-arrhythmic drug.

Exclusion Criteria:

1. Major valvular diseases needing surgical intervention.
2. Presence of a left atrial thrombus on recent imaging.
3. Recent myocardial infarction or severe heart failure (LVEF ≤ 30%).
4. Current Severe Infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from Atrial Arrhythmia Recurrence at 12 Months | 12 months after ablation procedure
  Proportion of participants free from atrial fibrillation/atrial flutter/atrial tachycardia recurrence at 12 months post-ablation.

SECONDARY OUTCOMES:
Procedural Safety | From enrollment to completion of follow-up（at least 12 months）
  Incidence of procedural complications such as esophageal injury and pulmonary vein stenosis.
Symptom Relief and Quality of Life Enhancement. | From enrollment to completion of follow-up（at least 12 months）
  Improvement in clinical symptoms (EHRA score) and quality of life measurements (Short Form 36 HealthSurvey).
Atrial Fibrillation Burden Reduction | From enrollment to completion of follow-up（at least 12 months）
  Reduction in atrial fibrillation burden assessed through follow-up evaluations.

CONTACTS AND LOCATIONS:
Locations (1):
- No. 241, West Huaihai Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP